CLINICAL TRIAL: NCT05741827
Title: YOUhealTH - a Study to Improve Cardiovascular Health in Adolescents and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VASCage GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: nC_FNA-0029_004
Record Dates: First submitted 2022-12-22; First posted 2023-02-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-07

CONDITIONS: Cardiovascular Diseases; Atherosclerosis
Keywords: Cardiovascular Risk Factors; Prevention; Diet; Physical Activity
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): Lifestyle intervention with focus on increased physical activity and healthy diet.
  Interventions: Behavioral: Lifestyle intervention
- Control group (No Intervention): No lifestyle intervention. No change in physical activity or diet.

INTERVENTIONS:
Behavioral: Lifestyle intervention — Lifestyle intervention focusing on diet and physical activity
  Arms: Interventional group

SUMMARY:
The goal of this single-center prospective randomized controlled parallel 2-arm intervention study is to test a lifestyle intervention focusing on diet and physical activity in students and at least one legal guardian to improve cardiovascular risk factor profiles.

The primary objective of this study ist to evaluate the efficacy of a health promotion intervention (intervention group) over the course of a year using a participative approach compared to a control group in 14- to 17-year-olds and at least one legal guardian.

Further study objectives are to determine the effect of the health promotion intervention on the change of the score of the individual health metric components, on the absolute health metric score, on the change in intima-media thickness and pulse-wave velocity and cardiovascular health (such as blood pressure, non-HDL-cholesterol, BMI) as well as health literacy with regards to CVDs, especially stroke, in both age-groups.

Furthermore, a biobank will be collected.

DETAILED DESCRIPTION:
YOUhealTH is a single-center prospective randomized controlled parallel 2-arm intervention study with the aim to test a lifestyle intervention focusing on diet and physical activity in students and at least one legal guardian to improve cardiovascular risk factor profiles. The lifestyle intervention is designed using a participative approach of adolescents who are part of the study team and design the intervention. This intervention is applied to students aged 14- to 17-years and at least one legal guardian for the duration of one year. At the beginning and the end of the intervention, an examination including a blood draw, a structured medical interview, anthropometrics including blood pressure measurement, ultrasonography of the aorta and the carotid artery, pulse-wave velocity and bioelectrical impedance measurement as well as FibroScan (a liver fat and elasticity measurement) is conducted and the effects of the intervention are evaluated compared to the control group receiving no intervention. Students and their legal guardians are randomized to the intervention or control group in a school-wise manner and in a 4:3 ratio.

The primary objective is to determine the effect of the health intervention with regards to the change of the health metric components diet and physical activity of the Life's Essential Eight score of the American Heart Association. Further study objectives are to evaluate the effect of the health promotion intervention on the change of the score of the individual health metric components, on the absolute health metric score, on the change in intima-media thickness and pulse-wave velocity and cardiovascular health (such as blood pressure, non-HDL-cholesterol, BMI) as well as health literacy with regards to CVDs, especially stroke, in both age-groups.

Furthermore, a long-term follow-up by means of record linkage is planned and a biobank will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents at the age of 14 to 17 years and at least one legal guardian willing to participate
* Signed informed consent of subjects and legal guardian

Exclusion Criteria:

* Persons, who are suspended upon a court order or upon other legal processes or are accommodated according to the Hospitalization Act, or for whom a custodian is appointed (or appointment is initiated).
* Persons with impaired power of judgment
* Persons who are currently engaged in military or community service
* Pregnancy of study participants

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Efficacy of health promotion intervention | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The efficacy of the health promotion intervention to improve cardiovascular health in 14- to 17 year-olds and at least one legal guardian measured by means of change of the "2022 cardiovascular health metrics score (0-100 points)" for the components of diet and physical activity from baseline to follow-up of the intervention group using a participative approach compared to a control-group.

SECONDARY OUTCOMES:
Health promotion intervention | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health promotion intervention on both the change and the absolute values of the "2022 cardiovascular health metrics score (0-100 points)" and its components in the whole study group and in adolescents and adults separately.
Health literacy | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health intervention on health literacy (measured by means of a CVD (HELMA; score) and stroke knowledge questionnaire (%)).
Pulse-wave velocity change | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health intervention on pulse-wave velocity (m/s)
Intima-media thickness change | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health intervention on intima-media thickness (µm).
Liver fat content change | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health intervention on liver fat content (dB/m).
Blood pressue change | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health intervention on blood pressure (mmHg).
Body-/fat composition change | Baseline visit until follow-up visit (at 12+/- 2 months)
  The effect of the health intervention on body-/fat composition (%)
Visceral fat thickness change | Baseline visit until follow-up visit (at 12+/- 2 months)
  The effect of the health intervention on abdominal visceral fat thickness (mm).
Physical activity change | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The effect of the health intervention on the average minutes of moderate to vigorous physical activity per day (min/day).
Risk profile - e.g. blood lipids | Baseline visit until follow-up visit (at 12 +/- 2 months)
  Risk profiles (e.g. blood lipids such as LDL-C (mg/dl)) of adolescents will be compared to their legal guardian(s).
Risk profile - e.g. Blood sugar | Baseline visit until follow-up visit (at 12+/- 2 months)
  Risk profiles (e.g. blood sugar (HbA1c (%)) of adolescents will be compared to their legal guardian(s).
Risk profile - Healthy diet | Baseline visit until follow-up visit (at 12+/- 2 months)
  Risk profiles (healty diet (MEPA score;%)) of adolescents will be compared to their legal guardian(s).
Risk profile - Smoking | Baseline visit until follow-up visit (at 12+/- 2 months)
  Risk profiles (smoking (questionnaire, score) of adolescents will be compared to their legal guardian(s).
Cardiovascular risk factor description - hypertension | Baseline visit until follow-up visit (at 12 +/- 2 months)
  The prevalence of traditional cardiovascular risk factors such as hypertension (mmHg) in the Tyrolean youth and their legal guardians will be described.
Cardiovascular risk factor description - obesity | Baseline visit until follow-up visit (at 12+/- 2 months)
  The prevalence of traditional cardiovascular risk factors such as obesity (e.g.BMI (kg/m^2)) in the Tyrolean youth and their legal guardians will be described.
Cardiovascular risk factor description - dislipidemia | Baseline visit until follow-up visit (at 12+/- 2 months)
  The prevalence of traditional cardiovascular risk factors such as dyslipidemia (e.g. LDL-C (mg/dl)) in the Tyrolean youth and their legal guardians will be described.
Cardiovascular risk factor description - diabetes | Baseline visit until follow-up visit (at 12+/- 2 months)
  The prevalence of traditional cardiovascular risk factors such as diabetes (HbA1c (%)) in the Tyrolean youth and their legal guardians will be described.
Lifestyle factor description - unhealthy diet | Baseline visit until follow-up visit (at 12+/- 2 months)
  The prevalence of lifestyle factors such as unhealthy diet (MEPA-score; %) in the Tyrolean youth and their legal guardians will be described.
Lifestyle factor description - sedentary lifestyle | Baseline visit until follow-up visit (at 12+/- 2 months)
  The prevalence of lifestyle factors such as sedentary lifestyle (Physical activity component of of Life's Essential 8 assessment; %) in the Tyrolean youth and their legal guardians will be described.
Lifestyle factor description - smoking | Baseline visit until follow-up visit (at 12+/- 2 months)
  The prevalence of lifestyle factors such as smoking (YES/NO, cigarettes per day) in the Tyrolean youth and their legal guardians will be described.
High-risk population exploration | Baseline visit until follow-up visit (at 12+/- 2 months)
  High-risk populations (Life's essential 8 score; %) based on school type, age, sex and region of residence will be explored.
Time trends | Baseline visit until follow-up visit (at 12+/- 2 months)
  Time trends in risk-profiles will be evaluated by comparison to the data from the "Early vascular Ageing" and the "Early Vascular Ageing in YOUth" study.
Long-term Intervention - CVD events | Every 2-5 years, on average for the duration of 50 years
  Evaluation of predictors for later cardio- and cerebrovascular disease (events or deaths) in adolescents and their legal guardian by record linkage to electronic health record.
Long-term Intervention - any deaths | Every 2-5 years, on average for the duration of 50 years
  Evaluation of predictors for later mortality in adolescents and their legal guardian by record linkage to death registry.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Knoflach, Assoc.-Prof., Principal Investigator — Medical University of Innsbruck
Locations (1):
- Department for Neurology, Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No